CLINICAL TRIAL: NCT01685515
Title: Phase 1 Study of Oral Decitabine and Tetrahydrouridine (THU) in Patients With High Risk Sickle Cell Disease
Brief Title: Study of Decitabine and Tetrahydrouridine (THU) in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yogen Saunthararajah (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Yogen Saunthararajah, Staff in the Department of Hematology and Oncology, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASE 10Z11
Record Dates: First submitted 2012-09-06; First posted 2012-09-14 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Decitabine; Tetrahydrouridine; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Decitabine and Tetrahydrouridine (Experimental): Oral Decitabine and Tetrahydrouridine
  Interventions: Drug: Oral Decitabine and Tetrahydrouridine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Decitabine and Tetrahydrouridine — Oral Decitabine and Oral Tetrahydrouridine (THU) given 1-2 hours apart on 2 consecutive days over 8 weeks
  Other Names: Dacogen, 5-aza-2'-deoxycytydine, THU
  Arms: Oral Decitabine and Tetrahydrouridine
Drug: Placebo — Plain water will be dispensed at a similar volume and in the same containers as study drug. The water placebo has a similar appearance and taste to the study drug, since the study drug is highly diluted in water.
  Other Names: Water
  Arms: Placebo

SUMMARY:
The purposes of this study are to observe if oral tetrahydrouridine and decitabine can increase fetal hemoglobin levels and improve the symptoms of sickle cell disease, and to monitor how patient's bodies react to oral tetrahydrouridine and decitabine.

DETAILED DESCRIPTION:
The purposes of this study are to observe if oral tetrahydrouridine and decitabine can increase fetal hemoglobin levels and improve the symptoms of sickle cell disease, and to monitor how patient's bodies react to oral tetrahydrouridine and decitabine. The overall purpose is to develop disease modifying treatment for sickle cell disease that is less cytotoxic than the current standard of care, and which can directly and more efficiently reactivate fetal hemoglobin levels. The hypothesis is that patients treated with oral tetrahydrouridine and decitabine will have the same chance of severe non-hematologic toxicities as the placebo group. The primary end-point is ≥ grade 3 non-hematologic toxicity. The investigators' hypothesis is that patients in the treatment groups receiving oral THU-decitabine 2X/week over 8 weeks (n=15) will be equivalent to placebo group (n=10) with regards to the chance of ≥ grade 3 non-hematologic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Written, informed consent provided by the subject before study entry.
* Confirmed Sickle Cell Disease (SCD) (SS, S-b0-thalassemia, S-b+-thalassemia or SC on hemoglobin electrophoresis).
* Symptomatic SCD while on 6 months of HU OR symptomatic SCD and intolerant of HU (unable or unwilling to take HU due to hematological or other toxicities). Symptomatic SCD is defined as having one of following:

  * Fetal Hemoglobin (HbF) <5%, OR
  * 3 or more pain episodes per year requiring parenteral narcotics, OR
  * 1 or more acute chest syndrome episodes, OR
  * Hemoglobin <9 g/dL and absolute reticulocyte count <250,000/mm3.
* Subject is in his/her steady state and not amidst any acute complication due to SCD (i.e., hospitalization, acute pain, or acute chest syndrome in the past 14 days).
* Regular compliance with comprehensive care and previous therapy.

Exclusion Criteria:

* Inability to give informed consent.
* Experienced severe sepsis or septic shock within the previous 12 weeks.
* Last HU dose was ingested within the previous 4 weeks.
* Currently pregnant or breast-feeding.
* Alanine aminotransferase (ALT) greater than or equal to two times (2X) the upper limit of normal or albumin <2.0 mg/dL or direct (conjugated) bilirubin greater than or equal to 1.5 mg/dl.
* Serum creatinine >2.9 mg/dL and calculated creatinine clearance <30 mL/min.
* Platelet count >800 x 109/L.
* Absolute neutrophil count <1.5 x 109/L.
* Female of active childbearing potential who is unwilling to use at least one of the two following forms of birth control:

  (i) not having heterosexual sexual contact beginning at the screening visit and continuing until 4 weeks after the last dose of THU-decitabine OR (ii) intrauterine device (IUD).
* Sexually active male who is unwilling to use a condom when engaging in any sexual contact with a female with child-bearing potential, beginning at the screening visit and continuing until 4 weeks after taking the last dose of THU-decitabine. This requirement applies also to males who have had a successful vasectomy.
* Altered mental status or recurrent seizures requiring anti-seizure medications.
* Moribund or any concurrent disease (e.g., hepatic, renal, cardiac, metabolic) of such severity that death within 24 weeks is likely.
* Concurrent diagnosis of malignancy including myelodysplastic syndromes (MDS), leukemia, or an abnormal karyotype.
* Vitamin-B12, folate, or iron deficient (until corrected).
* New York Heart Association (NYHA) class III/IV status.
* Eastern Co-operative Oncology Group (ECOG) performance status greater than or equal to 3.
* Participant is on chronic transfusion therapy (e.g., for history of Transient Ischemic Attack (TIA) or stroke) and medically contraindicated to discontinue transfusions (unless multiple allo-antibodies prevent the patient from getting transfusions as scheduled).
* Known history of illicit drug or alcohol abuse within the past 12 months.
* Other experimental or investigational drug therapy in the past 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Non-hematologic toxicity | 12 weeks
  Toxicities will be evaluated on a weekly basis and will be classified according to their grade and relationship to study treatment. Chi-square testing will be employed to examine the difference in number of patients with grade 3 or greater non-hematologic toxicity between treatment and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yogen Saunthararajah, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Molokie R, Lavelle D, Gowhari M, Pacini M, Krauz L, Hassan J, Ibanez V, Ruiz MA, Ng KP, Woost P, Radivoyevitch T, Pacelli D, Fada S, Rump M, Hsieh M, Tisdale JF, Jacobberger J, Phelps M, Engel JD, Saraf S, Hsu LL, Gordeuk V, DeSimone J, Saunthararajah Y. Oral tetrahydrouridine and decitabine for non-cytotoxic epigenetic gene regulation in sickle cell disease: A randomized phase 1 study. PLoS Med. 2017 Sep 7;14(9):e1002382. doi: 10.1371/journal.pmed.1002382. eCollection 2017 Sep. PMID 28880867